CLINICAL TRIAL: NCT05418127
Title: A Randomized, Double-blinded, Placebo-controlled, Parallel Study, to Assess the Effect of Traditionally Fermented Organic Coconut Milk Kefir on Gastrointestinal Symptoms in Healthy Adults
Brief Title: An Efficacy Trial in the Research Area of Gastrointestinal Health & Bloating
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coconut Goodness Food Products Inc. (Industry)
Responsible Party: Principal Investigator, Linda Peers, Principal Investigator, Coconut Goodness Food Products Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-151
Record Dates: First submitted 2022-06-01; First posted 2022-06-14 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Gastrointestinal Dysfunction
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, parallel study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only one representative of sponsor and two Atlantia Clinical Trials representatives are unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 Participants receiving Placebo product. (Placebo Comparator): Solution of filtered water, Calcium Carbonate powder, and coconut extract.
  Interventions: Other: Placebo
- 30 Participants receiving Active product. (Active Comparator): Traditionally-fermented coconut milk kefir.
  Interventions: Dietary Supplement: Active

INTERVENTIONS:
Dietary Supplement: Active — Traditionally-fermented coconut milk kefir
  Arms: 30 Participants receiving Active product.
Other: Placebo — Solution of Calcium Carbonate and coconut extract
  Arms: 30 Participants receiving Placebo product.

SUMMARY:
A randomized, double-blinded, placebo-controlled, parallel study, to evaluate the effect of 8-week supplementation of a traditionally fermented organic coconut milk kefir compared to placebo on gastrointestinal symptoms in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study and comply with its procedures, including but not limited to consuming study product, adhering to visit schedule and e-diary/questionnaires, abstaining from products outlined in Section 5.8 of Study Protocol.
2. Able and willing to give written informed consent.
3. Adults aged between 25 to 54 years, inclusive.
4. Self-reported bloating on at least 3 occasions over the 7-day period immediately prior to enrolment (confirmed by selecting any option other than 'None' in response to the daily electronic diary Bloating question in the electronic diary questionnaire completed prior to enrolment).

Exclusion Criteria:

1. Participants who are pregnant or wish to become pregnant during the trial.
2. Participants who are lactating and/or currently breastfeeding.
3. Participants currently of childbearing potential, but not using an effective method of contraception for at least 30 days prior to dosing, as outlined below:

   1. Complete abstinence from intercourse prior to administration of the study product, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study product in cases where participant discontinues the trial prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit).
   2. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that participant.
   3. Sexual partner(s) is/are exclusively female.
   4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g. male condom, female diaphragm), or contraceptive pill/patch/injection/ring. The participant must be using this method for at least 30 days prior to and 2 weeks following the end of the trial.
   5. Use of any intrauterine device (IUD) or contraceptive implant. The participant must have the device inserted at least 30 days prior to the first Screening Visit, throughout the trial, and 2 weeks following the end of the trial.
4. Participants who have a history of histamine intolerance (i.e., intolerance to fermented food) or any known coconut or tree nut allergy.
5. Participants who have consumed prebiotic or probiotic supplements in the 14 days prior to screening (Visit 1).
6. Participants have consumed fermented coconut/kefir products in the 14 days prior to screening (Visit 1) and are intending to consume such products during the course of the trial.
7. Participants who have used oral antibiotics in the 90 days prior to screening (Visit 1).
8. Participants who have had gastrointestinal surgery (e.g., colectomy, gall bladder removal, gastric bypass) - appendectomy not considered an exclusionary surgery.
9. Participants who have any significant health conditions or current medications that would prevent them from fulfilling the trial requirements, put the Participant at risk or would confound the interpretation of the trial results as judged by the investigator on the basis of medical history, medication history, and routine laboratory test results.
10. Participants who cannot safety stop taking prescription medication for the duration of the trial
11. Participants may not be receiving treatment involving experimental drugs. If the Participant has been in a recent experimental trial, these must have been completed not less than 60 days prior to screening (Visit 1).
12. Participants who have used any immunosuppressant or chemotherapy medications, including marcaptopurine, azothioprine, or methotrexate in the last 5 years.
13. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
14. Any Participant who is an employee of the investigational site or an Atlantia Clinical Trials employee or their close family member or a member of their household.

Ages: 25 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of Participants who report a change in the maximum severity of their bloating in a daily eDiary. | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention the effect of 8-week supplementation of a fermented coconut milk kefir compared to Placebo on the severity of bloating from baseline to Week 8 (confirmed by selecting a lower category of severity of bloating during the 7-day period prior to end of intervention compared to the 7-day period prior to Baseline on the day with their worst symptom rating).

SECONDARY OUTCOMES:
Change in mean daily severity of Abdominal Pain symptoms of Participants (as recorded in the daily e-diary Abdominal Pain question). | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention the effect of 8-week supplementation of a fermented coconut milk kefir compared to Placebo on the severity of abdominal pain (as recorded in the daily e-diary Abdominal Pain question) during the 7-day period prior Baseline compared to the 7-day period prior to end of intervention.
Change in mean daily severity of Abdominal Discomfort symptoms of Participants (as recorded in the daily e-diary Abdominal Pain question). | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention the effect of 8-week supplementation of a fermented coconut milk kefir compared to Placebo on the severity of abdominal discomfort (as recorded in the daily e-diary Abdominal Discomfort question) during the 7-day period prior Baseline compared to the 7-day period prior to end of intervention.
Change in proportion of Participants experiencing Flatulence/Gas symptoms (selecting any option other than 'None' in response to the daily e-diary Flatulence/Gas question). | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention the effect of 8-week supplementation of a fermented coconut milk kefir compared to Placebo on the severity of flatulence/gas (confirmed by selecting any option other than 'None' in response to the daily e-diary Flatulence/Gas question) during the 7-day period prior Baseline compared to the 7-day period prior to end of intervention.
Difference between product groups of self-reported symptom improvement from the Global Impression of Change Scale at end of intervention. | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention the effect of 8-week supplementation of a fermented coconut milk kefir compared to Placebo on their overall perception of their bloating symptoms as reported in a product satisfaction questionnaire at week 8. Subjects rate perception of change in bloating using a visual analogue scale (VAS) rated from "There has been no change to my bloating" to "There has been a significant change to my bloating"

OTHER OUTCOMES:
Change in Hs-CRP | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention the effect of 8-week supplementation of a fermented coconut milk kefir compared to Placebo on Hs-CRP from baseline to Week 8.
Change in microbiome profile | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention the effect of 8-week supplementation of a fermented coconut milk kefir compared to Placebo on Change in microbiome profile from baseline to Week 8.
Overall product satisfaction questionnaire as measured by the Overall Product Satisfaction Questionnaire | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention their overall product satisfaction following an 8-week supplementation of a fermented coconut milk kefir compared to Placebo. Questions about the taste, ease of us and desire to continue use are answered using visual analogue scales (VAS) (e.g., 'I like it very much' -> 'I do not like it at all')
Change in quality of life assessed by the Short Form-36 (SF-36) | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention the effect of 8-week supplementation of a fermented coconut milk kefir compared to Placebo on Participant Quality of Life from baseline to Week 8 using the SF-36. The SF-36 is a self-administered questionnaire comprising 36-items measuring eight health domains: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health (5 items).
Change in daily performance (energy and mental clarity) assessed daily eDiary | 8 weeks
  To evaluate in healthy adults who experience gastrointestinal bloating or distention the effect of 8-week supplementation of a fermented coconut milk kefir compared to Placebo on daily performance (energy and mental clarity) reported in daily eDiary. Questions about energy and mental clarity over the previous 24 hours will be answered on a 5 point scale from strongly disagree to strongly agree.
Incidence of Adverse Events (AEs) [Safety] | 8 weeks
  To evaluate incidence of AEs in participants supplemented with a fermented coconut milk kefir compared to Placebo
Incidence of mild, moderate, and severe AEs [Safety] | 8 weeks
  To evaluate incidence of mild, moderate, and severe AEs in participants supplemented with a fermented coconut milk kefir compared to Placebo
Incidence of AEs by MEDRA System Organ Classification (SOC) and preferred term (PT) [Safety] | 8 weeks
  To evaluateof AEs by MEDRA System Organ Classification (SOC) and preferred term (PT) in participants supplemented with a fermented coconut milk kefir compared to Placebo
Incidence of Vital Parameter AEs [Safety] | 8 weeks
  To evaluate incidence vital parameter (blood pressure, heart rate, temperature) AEs in participants supplemented with a fermented coconut milk kefir compared to Placebo
Incidence of Serious Adverse Events (SAEs) [Safety] | 8 weeks
  To evaluate incidence of SAEs in participants supplemented with a fermented coconut milk kefir compared to Placebo

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Boetto, FNP-C, Principal Investigator — Atlantia Clinical Trials Ltd.
Locations (1):
- Atlantia Clinical Trials Ltd., Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Those conducting research in the area of Gastrointestinal Health & Bloating